CLINICAL TRIAL: NCT07101458
Title: Feasibility and Acceptability of the Promoting Resilience in Stress Management (PRISM) Intervention Among Adolescents (10 - 19 Years) Living With HIV in Eswatini: A Single Site, Single-Blind, Randomized Controlled Pilot Clinical Trial
Brief Title: The Eswatini PRISM Study on Adolescents Living With HIV
Acronym: PRISM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eswatini Nazarene Health Institutions (Other)
Collaborators: Baylor Foundation Eswatini (Unknown); Dana-Farber Cancer Institute (Other); University of Eswatini (Unknown)
Responsible Party: Principal Investigator, Musa Lewis Nhlabatsi, Family Nurse Practitioner, Eswatini Nazarene Health Institutions
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EHHRRB 075/2025
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-07

CONDITIONS: Human Immunodeficiency Virus; Psychological Stress
Keywords: Adolescents; Health-related quality of life; Human immunodeficiency virus; Psychological distress; Promoting Resilience in Stress Management; Resilience
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Single-site, single-blind, parallel randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Promoting Resilience in Stress Management (PRISM)
  Individual, 1:1 version of the Promoting Resilience in Stress Management intervention.
  Interventions: Behavioral: Promoting Resilience in Stress Management intervention
- Standard Psychosocial Care (No Intervention): Standard psychosocial care includes comprehensive psychosocial evaluations and referrals to behavioural health services, financial assistance, and various social support resources available at the health facility.

INTERVENTIONS:
Behavioral: Promoting Resilience in Stress Management intervention — PRISM is a manualized, skills-based training program comprised of three 60-minute, one-on-one sessions designed to build resilience resources (stress management, goal-setting, cognitive-reframing, and meaning-making) in adolescents and young adults (AYAs). The sessions are scheduled every 1-2 weeks based on participant preference. In this study, the PRISM sessions will be facilitated by trained nurses who hold bachelor's degrees in Nursing Science with a specialisation in mental health.
  Other Names: PRISM; PRISM intervention; PRISM program
  Arms: Treatment Arm

SUMMARY:
Adolescents living with Human Immunodeficiency Virus (ALHIV) are at an increased risk of experiencing psychological distress and adverse mental health outcomes, particularly in low- to middle-income countries (LMICs). Although interventions aimed at promoting resilience have demonstrated potential in enhancing psychosocial outcomes among adolescents with chronic illnesses in high-income settings, there is a paucity of evidence from LMICs. This study protocol aims to outline a comprehensive framework for evaluating the feasibility, acceptability, and effectiveness of the Promoting Resilience in Stress Management (PRISM) intervention in comparison to standard psychosocial care among ALHIV in a LMIC, such as Eswatini (formerly known as Swaziland). Additionally, it seeks to gather qualitative insights from both participants and PRISM coaches regarding the PRISM program. Exploratory outcomes under investigation are psychological distress, resilience, and HIV health-related quality of life. We hypothesise that:

1. Participants in the PRISM intervention group will experience reduced psychological distress compared to those in the control arm.
2. Participants in the PRISM intervention group will report improved HIV health-related quality of life after receiving the intervention compared to the control group.
3. Participants in the intervention arm will have higher resilience scores after receiving the intervention compared to those receiving usual psychosocial care.

DETAILED DESCRIPTION:
This study employs an explanatory sequential mixed-methods design to rigorously evaluate the Promoting Resilience in Stress Management (PRISM) intervention. In the initial quantitative phase, a single-site, single-blind, pilot randomized controlled trial (RCT) will be conducted. A sample of (n=140) ALHIV will be recruited and randomly assigned to either the PRISM intervention arm or a control arm receiving standard psychosocial care. The PRISM intervention, a manualized, skills-based training program, originally comprises six 30-60-minute, one-on-one sessions designed to enhance resilience resources, including stress management, goal-setting, cognitive reframing, and meaning-making, in adolescents and young adults (AYAs). For the purposes of this trial, the PRISM intervention will be adapted to consist of three 60-minute sessions, delivered at intervals of 1-2 weeks based on participant preference. Participants in both arms will complete validated survey instruments to assess exploratory outcomes, including psychological distress, resilience, and HIV-related quality of life. Data collection will occur at baseline (T0), and at 3 months (T1), 6 months (T2), 9 months (T3), and 12 months (T4) post-enrollment. The researchers will then evaluate the feasibility, acceptability, and effectiveness of the PRISM intervention based on these outcomes.

In the second phase of the study, an Exploratory-Descriptive Qualitative (EDQ) research design will be employed to investigate the experiences and perceptions of participants engaged in the PRISM program. Data collection will involve the use of semi-structured interview guides administered to nurse PRISM coaches and a purposively selected sample of ALHIV from the intervention arm of the pilot clinical trial. The collected data will undergo rigorous thematic analysis to elucidate key insights into the participants' experiences and perceptions of the PRISM intervention, thereby contributing to a deeper understanding of its implementation and impact.

ELIGIBILITY:
Inclusion Criteria for the Clinical Trial:

* Adolescents living with HIV aged 10-19 years.
* Adolescents living with HIV who are cognitively able to participate in interviews (based on their medical history).
* Adolescents living with HIV who will have a score > 13 on the Kessler Screening Scale for Psychological Distress (K6).

Exclusion Criteria for the Clinical Trial:

* Adolescents who refuse to participate.
* Adolescents whose parents/caretakers (for <18 years) will not consent to their participation.
* Adolescents who will report having suicidal thoughts (i.e., who will respond yes to one item asking if they thought of killing themselves in the last 30days). This exclusion is based on the understanding that the PRISM intervention was not designed to address suicidal ideation, as confirmed by its developers. Such individuals will be referred to a licensed psychologist following the study's established referral plan, thereby ensuring they receive the appropriate care and support.

Inclusion criteria for a support person:

The PRISM intervention requires a caretaker or parent to be invited by the study participant to join the third session.

• Parent or caretaker should be ≥ 18 years of age and consent to participation.

Exclusion criteria for a support person:

• A parent or caretaker who refuses to participate.

Eligibility Criteria for Participation in Semi-Structured Interviews Post Intervention

Inclusion criteria for participants:

* Adolescents who have been in the treatment arm of the PRISM intervention pilot clinical trial.
* Adolescents who completed all sessions of the PRISM intervention.
* Adolescents who are willing to be audio taped.

Exclusion criteria for participants:

• Participants who meet the inclusion criteria but are unwilling to provide informed consent or assent and/or parental consent.

Inclusion criteria for implementers:

• PRISM coaches who offered all sessions of the PRISM intervention and who will be willing to be audio-taped.

Exclusion criteria for implementers:

• PRISM coaches who meet the inclusion criteria but are unwilling to provide informed consent to participate.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the PRISM intervention | 12 months outcome assessment point.
  Feasibility of the PRISM intervention will be defined as priori >70% program completion of the three PRISM sessions among enrolled participants.
Acceptability of the PRISM | 12 months outcome assessment point.
  Acceptability of the PRISM intervention, which is a primary outcome, will be measured using the Client Satisfaction Questionnaire (CSQ-8), an 8-item measuring participant's opinions and assessments of the intervention. Each item is rated on a 4-point Likert scale, where responses range from 1 (indicating dissatisfaction) to 4 (indicating high satisfaction). The total score, which ranges from 8 to 32, is derived by summing the responses to all eight items. A higher score on the CSQ-8 reflects greater satisfaction with the PRISM intervention.

SECONDARY OUTCOMES:
Effectiveness of the PRISM intervention | At 12 months outcome assessment point.
  Effectiveness of the PRISM intervention will be determined by comparing the changes in psychological distress, resilience and HIV health-related quality of life mean scores pre- and post-intervention for both the treatment and usual care groups of the trial. A statistically significant reduction in mean scores of the above-mentioned outcomes in the treatment group compared to the control group will suggest that the PRISM intervention is effective.
Psychological distress | At 3, 6, 9, and 12-months outcome assessment points.
  Psychological distress will be assessed by the Kessler Psychological Distress Scale (K6), a self-administered screening tool developed to screen for non-specific psychological distress and serious mental illness in various populations. Participants will be asked to rate how often they experienced symptoms in the past thirty days using the K6 questionnaire. They will rate their experiences on a 5-point Likert scale for each question, where 0 = none of the time, 1 = a little of the time, 2 = some of the time, 3 = most of the time, and 4 = all of the time. A total score of psychological distress will be computed by summing the scores for all six items. The K6 questionnaire has a total score ranging from 0 to 24 points, with higher scores indicating severe psychological distress.
Resilience | At 3, 6, 9, and 12-months outcome assessment points.
  Resilience will be assessed with the Connor-Davidson Resilience Scale 10-Item (CD-RISC 10). The CD-RISC 10 consists of 10 items, and respondents rate each item on a 5-point Likert scale, ranging from 0 (not true at all) to 4 (true nearly all the time). The total score for the CD-RISC 10 ranges from 0 to 40, with higher scores indicating greater resilience.
HIV health-related quality of life | At 3, 6, 9, and 12-months outcome assessment points.
  The HIV health-related quality of life of adolescents living with HIV will be assessed using the World Health Organization Quality of Life Instrument-HIV (WHOQOL-HIV). Each item within the WHOQOL HIV BREF instrument is rated on a 5-point scale: 1 = not at all, 2 = a little, 3 = a moderate amount, 4 = very much, and 5 = an extreme amount. Participants in the study will score how they perceive the five domain items in the WHOQOL targeting HIV. An average score from each domain will be computed to have a total health quality of life for each participant. Then, higher scores reflect higher satisfaction or better functioning in these domains, suggesting a better overall quality of life.

OTHER OUTCOMES:
Experiences and perceptions of ALHIV and PRISM coaches regarding the PRISM intervention. | Within a month after completing the intervention.
  In-depth, face-to-face interviews will be conducted with nurse PRISM coaches and conveniently selected ALHIV participants in the intervention arm of the pilot clinical trial using a semi-structured interview guide.

CONTACTS AND LOCATIONS:
Overall Officials: Musa L. Nhlabatsi, MSc, Principal Investigator — Eswatini Nazarene Health Institutions; Mduduzi C. Shongwe, PhD, Study Director — Department of Midwifery Science, University of Eswatini; Debrah Vambe, MD, Study Director — Baylor Foundation Eswatini; Kay Alexander, MD, Study Director — Baylor Foundation Eswatini; Nobuhle Mthethwa, MPH, Study Director — Eswatini Ministry of Health (MOH)/Eswatini National Health AIDS; Joyce Yi-Frazier, PhD, Study Director — Dana-Farber Cancer Institute (DFCI)
Locations (1):
- Raleigh Fitkin Memorial Hospital-Baylor College of Medicine Children's Foundation Clinic, Manzini, Manzini Region, Eswatini

IPD SHARING:
Plan to Share IPD: Yes
De-identified data generated from this study will be securely uploaded to a dedicated Baylor Foundation Eswatini data server repository to facilitate data sharing in accordance with the foundation's data management policy. The study protocol and statistical analysis plan will be publicly accessible on ClinicalTrials.gov, in compliance with federal regulations or as stipulated by the conditions of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 6 months after publication for 10 years.
Access Criteria: Anonymized participant data will be shared with the scientific community according to the Baylor Foundation Eswatini data sharing policy upon request.

REFERENCES:
- [Background] Rosenberg AR, Zhou C, Bradford MC, Salsman JM, Sexton K, O'Daffer A, Yi-Frazier JP. Assessment of the Promoting Resilience in Stress Management Intervention for Adolescent and Young Adult Survivors of Cancer at 2 Years: Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2021 Nov 1;4(11):e2136039. doi: 10.1001/jamanetworkopen.2021.36039. PMID 34817581
- [Background] Rosenberg AR, Bradford MC, McCauley E, Curtis JR, Wolfe J, Baker KS, Yi-Frazier JP. Promoting resilience in adolescents and young adults with cancer: Results from the PRISM randomized controlled trial. Cancer. 2018 Oct 1;124(19):3909-3917. doi: 10.1002/cncr.31666. Epub 2018 Sep 19. PMID 30230531
- [Background] Rosenberg AR, Yi-Frazier JP, Eaton L, Wharton C, Cochrane K, Pihoker C, Baker KS, McCauley E. Promoting Resilience in Stress Management: A Pilot Study of a Novel Resilience-Promoting Intervention for Adolescents and Young Adults With Serious Illness. J Pediatr Psychol. 2015 Oct;40(9):992-9. doi: 10.1093/jpepsy/jsv004. Epub 2015 Feb 11. PMID 25678533
- [Background] Yi-Frazier JP, Hilliard ME, O'Donnell MB, Zhou C, Ellisor BM, Garcia Perez S, Duran B, Rojas Y, Malik FS, DeSalvo DJ, Pihoker C, Bradford MC, Scott S, Devaraj S, Rosenberg AR. Promoting Resilience in Stress Management for Adolescents With Type 1 Diabetes: A Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2428287. doi: 10.1001/jamanetworkopen.2024.28287. PMID 39158914